CLINICAL TRIAL: NCT02090933
Title: Clinical Protocol for an Open Label Study of Celecoxib (SC-58635) on the Acute Effect of Human UV-Irradiation
Brief Title: Celecoxib in Decreasing the Damaging Effects of Sunburn in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2014-00524; NCI-2014-00524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RSRB#10077 (Other: University of Rochester); N01-CN-85183-Step-1-Ext (Other: DCP); N01CN85183 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: No Evidence of Disease
MeSH Terms: interventions — Celecoxib; Ultraviolet Therapy

ARMS (1):
- Treatment (celecoxib) (Experimental): Participants undergo UV-irradiation to the right buttock at baseline, receive celecoxib PO BID for 10 days, and then undergo UV-irradiation to the left buttock.
  Interventions: Drug: Celecoxib; Other: Laboratory Biomarker Analysis; Procedure: UV Light Therapy

INTERVENTIONS:
Drug: Celecoxib — Given PO
  Other Names: SC-58635
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: UV Light Therapy — Undergo UV-irradiation
  Other Names: Light Therapy, UV; Therapy, UV Light; Ultraviolet Radiation Therapy

SUMMARY:
This clinical trial studies celecoxib in decreasing the damaging effects of sunburn in healthy volunteers. Celecoxib may reduce skin damage by blocking enzymes associated with sunburn in healthy volunteers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Quantify changes in the erythema response in human subjects exposed to a range of erythemic doses of solar-simulated ultraviolet light before and after celecoxib treatment.

II. Collect blood for genetic analysis of markers likely to modulate erythema response. This includes cyclooxygenase (COX), prostaglandin receptor, P53 and excision-repair polymorphisms.

OUTLINE:

Participants undergo ultraviolet (UV)-irradiation to the right buttock at baseline, receive celecoxib orally (PO) twice daily (BID) for 10 days, and then undergo UV-irradiation to the left buttock. Chromameter readings are obtained 24 hours post UV-irradiation.

ELIGIBILITY:
Inclusion Criteria:

* The subject has Fitzpatrick skin type I, II, or III
* If the subject is female and of childbearing potential (women are considered not of childbearing potential if they are at least 2 years post-menopausal and/or surgically sterile):

  * Has been using adequate contraception (e.g., condom, intrauterine device [IUD], diaphragm and spermicide gel combination) since her last menses and will use adequate contraception during the study, and
  * Is not lactating, and
  * Will begin taking study drug beginning 2 days after onset of menses
* The subject is willing to abstain from the use of other non-steroidal anti-inflammatory drugs (NSAIDs) for the duration of the study
* The subject is willing to abstain from the use of all topical agents applied to the buttocks for the duration of the study with the exception of lotion
* The subject is willing to participate for the duration of the study
* The subject has provided written informed consent prior to administration of any study related procedures

Exclusion Criteria:

* The subject is currently taking any medication that may alter the sunlight response or cause an adverse reaction
* The subject has a history of melanoma, lupus, psoriasis, rosacea, porphyria, photosensitivity disorder, connective tissue disorder, or any disease that would increase the risk associated with study participation
* The study has excessive hair, blemishes, nevi, uneven pigmentation, sunburn or suntan on the buttocks
* The subject has sun bathed or used a tanning bed to expose the buttocks within 12 months of admission to the study
* The subject has inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), a chronic or acute renal or hepatic disorder or a significant coagulation defect or any other condition which in the Investigator's opinion might preclude use of an NSAID (e.g., congestive heart failure)
* The subject has an active malignancy of any type; subjects who have a history of nonmelanoma skin cancer and have been treated are acceptable; subjects with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years prior to study enrollment are also acceptable
* The subject has active or suspected peptic ulceration or gastrointestinal bleeding
* The subject has received any investigational medication within 30 days prior to the first dose of study medication or is scheduled to receive an investigational drug other than celecoxib during the course of this study
* The subject has a known hypersensitivity to cyclooxygenase-2 inhibitors, sulfonamides, or NSAIDs
* The subject has significant medical or psychosocial problems that would make the subject a poor candidate, in the opinion of the principal investigator
* The subject is currently taking celecoxib

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-03; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Changes in the erythema response in human subjects exposed to a range of erythemic doses of solar-simulated ultraviolet light before and after celecoxib treatment | Baseline up to day 11

CONTACTS AND LOCATIONS:
Overall Officials: Alice Pentland, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States